CLINICAL TRIAL: NCT05912101
Title: Comparison of the Effects of Pericapsular Nerve Group (PENG), Suprainguinal Fascia Iliaca Compartment (S-FICB) and 3-1 Blocks on Comfort in Positioning for Unilateral Spinal Anesthesia and Postoperative Pain in Hip Fracture Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bozyaka Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022/49 ArdaTez
Record Dates: First submitted 2023-06-11; First posted 2023-06-22 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-06

CONDITIONS: Hip Fractures; Pain Management; Pain Postoperative; Spinal Anesthesia; Nerve Block/Methods
Keywords: Hip Fracture; Unilateral Spinal Anesthesia; Pericapsular Nerve Group Block; 3-1 Block; Suprainguinal Fascia Iliaca Compartment Block; Pain Management
MeSH Terms: conditions — Hip Fractures; Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (PENG) (Experimental): A convex USG Probe (1-5 mHz) is placed transversely on the SIAS (Spina Iliaca Anterior Superior). The probe is then rotated 45 degrees and aligned with the pubic ramus. In this position, the iliopubic eminence, ilipsoas muscle-tendon, femoral artery and pectineus muscle are observed. A 100 mm 21G block needle (Stimuplex A®:B. Braun Melsungen AG, Japan) is inserted in-plane from lateral to medial to the musculofascial plane with the psoas tendon in front and the pubic ramus behind and the injection is performed.
  Interventions: Procedure: Pericapsular Nerve Group Block
- Group 2 (S-FICB) (Experimental): A linear USG probe (7-13 mHz) is placed parasagittal to obtain an image of the SIAS. The probe is then shifted medially to identify the fascia iliaca, iliac muscle, internal oblique muscle and deep circumflex iliac artery. A 50 mm 21G block needle (Stimuplex A®:B. Braun Melsungen AG, Japan) is advanced in-plane from caudal to cephalic and injected between the fascia iliaca and iliac muscle.
  Interventions: Procedure: Suprainguinal Fascia Compartment Block
- Group 3 (3-1) (Experimental): A linear USG probe (7-13 mHz) is placed at the level of the femoral fold and the femoral vein-arterial-nerve is visualized. The femoral nerve is located below the fascia iliaca. At this point, a 50 mm 21G block needle (Stimuplex A®:B. Braun Melsungen AG, Japan) is inserted in-plane from lateral to medial and injected lateral to the femoral nerve. After injection, pressure is applied distal to the needle entry site to spread the local anesthetic proximally in the nerve sheath.
  Interventions: Procedure: 3-1 Block

INTERVENTIONS:
Procedure: Pericapsular Nerve Group Block — A convex USG Probe (1-5 mHz) is placed transversely on the SIAS (Spina Iliaca Anterior Superior). The probe is then rotated 45 degrees and aligned with the pubic ramus. In this position, the iliopubic eminence, ilipsoas muscle-tendon, femoral artery and pectineus muscle are observed. A 100 mm 21G block needle (Stimuplex A®:B. Braun Melsungen AG, Japan) is inserted in-plane from lateral to medial to the musculofascial plane with the psoas tendon in front and the pubic ramus behind and the injection is performed.
  Arms: Group 1 (PENG)
Procedure: Suprainguinal Fascia Compartment Block — A linear USG probe (7-13 mHz) is placed parasagittal to obtain an image of the SIAS. The probe is then shifted medially to identify the fascia iliaca, iliac muscle, internal oblique muscle and deep circumflex iliac artery. A 50 mm 21G block needle (Stimuplex A®:B. Braun Melsungen AG, Japan) is advanced in-plane from caudal to cephalic and injected between the fascia iliaca and iliac muscle.
  Arms: Group 2 (S-FICB)
Procedure: 3-1 Block — A linear USG probe (7-13 mHz) is placed at the level of the femoral fold and the femoral vein-arterial-nerve is visualized. The femoral nerve is located below the fascia iliaca. At this point, a 50 mm 21G block needle (Stimuplex A®:B. Braun Melsungen AG, Japan) is inserted in-plane from lateral to medial and injected lateral to the femoral nerve. After injection, pressure is applied distal to the needle entry site to spread the local anesthetic proximally in the nerve sheath.
  Arms: Group 3 (3-1)

SUMMARY:
Hip fracture is a common cause of surgery, especially in elderly patients. Unilateral spinal anesthesia in hip fracture surgery can prevent the undesirable effects of spinal anesthesia due to sympathetic blockade.

However, severe pain in hip fracture patients limits the positioning required for unilateral spinal anesthesia. The sedation and analgesia required to position patients with fractured hip remains inferior may cause respiratory depression, hemodynamic instability or postoperative cognitive impairment, especially in elderly patients. Lower extremity peripheral blocks can be used preoperatively to minimize the use of sedatives that may be required during positioning and to provide effective and safe analgesia.

DETAILED DESCRIPTION:
In the study, one anesthesiologist (Anesthesiologist A) will perform the relevant peripheral blocks according to the groups to which the patients are randomized; the other anesthesiologist (Anesthesiologist B) will perform unilateral spinal anesthesia in all patients blinded to the peripheral blocks.

On the day of surgery, the patients will first be taken to the block application room and standard monitoring (ECG, pulse oximetry, noninvasive blood pressure) will be applied in the supine position. In the pre-block period, individual pain assessment will be performed with the Visual Analog Scale (VAS - 0 cm = no pain / 10 cm = unbearable pain) and recorded on the case report form. After the pain assessment, disinfection of the block area will be performed with 10% povidone iodine (Batidex) in accordance with surgical sterilization rules. After sterilization, the relevant peripheral block will be performed by Anesthesiologist A under USG guidance. Intermittent negative aspiration will be performed during all interventions to detect possible vascular puncture. All groups will receive 30 ml of local anesthetic solution containing 5 mcg/ml adrenaline and bupivacaine at 0.25% concentration.

Group 1 (PENG Block): Convex USG Probe (1-5 mHz) is placed transversely on SIAS (Spina Iliaca Anterior Superior). The probe is then rotated 45 degrees and aligned with the pubic ramus. In this position, the iliopubic eminence, ilipsoas muscle-tendon, femoral artery and pectineus muscle are observed. A 100 mm 21G block needle (Stimuplex A®:B. Braun Melsungen AG, Japan) is inserted in-plane from lateral to medial to the musculofascial plane with the psoas tendon in front and the pubic ramus behind and the injection is performed.

Group 2 (Suprainguinal Fascia Iliaca Compartment Block) : Linear USG Probe (7-13 mHz) is placed parasagittal to obtain an image of the SIAS. The probe is then shifted medially to identify the fascia iliaca, iliac muscle, internal oblique muscle and deep circumflex iliac artery. A 50 mm 21G block needle (Stimuplex A®:B. Braun Melsungen AG, Japan) is advanced in-plane from caudal to cephalic and injected between the fascia iliaca and iliac muscle.

Group 3 (3-1 Block) Linear USG Probe (7-13 mHz) is placed at the femoral fold and femoral vein-arterial-nerve is visualized. The femoral nerve is located below the fascia iliaca. At this point, a 50 mm 21G block needle (Stimuplex A®:B. Braun Melsungen AG, Japan) is inserted in-plane from lateral to medial and injected lateral to the femoral nerve. After injection, pressure is applied distal to the needle entry site to spread the local anesthetic proximally in the nerve sheath.

The VAS score of the patients will be reevaluated and recorded during positioning for unilateral spinal anesthesia 30 minutes after the block is performed. Patients with VAS > 3 will be administered sedoanalgesia with propofol - ketamine combination as rescue analgesia before spinal anesthesia and recorded in the case report form. (1 = need sedoanalgesia / 2 = no need sedoanalgesia) Unilateral spinal anesthesia will be administered by Anesthesiologist B after the patient is positioned so that the fractured hip remains at the bottom. The quality of the patient's position will be evaluated by Anesthesiologist B administering spinal anesthesia and recorded on the case report form (0 = inadequate, 1 = adequate, 2 = good, 3 = optimal) All patients will be routinely administered 1000 mg acetominophen 3x1 in the postoperative period.

All patients will be followed up in terms of VAS score and possible opioid requirement in the postoperative 24 hours and evaluated in terms of satisfaction with the procedure.

Patients will be monitored for 24 hours in terms of undesirable side effects and if signs of vascular puncture, hematoma, LA toxicity are observed, these events will be recorded in the case report form and serious adverse reactions will be reported.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* American Society of Anesthesiologists Physical Status Classification(ASA) I,II and III
* Fully oriented and able to cooperate
* Consented to participate in the study by signing the informed consent form
* Patients with hip fracture and planned unilateral surgery with spinal anesthesia

Exclusion Criteria:

* Patients under 18 years of age
* Refusal to participate
* American Society of Anesthesiologists Physical Status Classification(ASA) IV-V
* Non-cooperation
* Coagulopathy or thrombocytopenia
* Allergic to local anesthetics and analgesics
* Patients with anatomical abnormalities or active infection at the points of application

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Positional Pain in Unilateral Spinal Anesthesia | 30 minutes after the block is performed
  Pain in the pre-block period and during unilateral spinal anesthesia positioning after the block will be evaluated by VAS score.

SECONDARY OUTCOMES:
Position Quality in Unilateral Spinal Anesthesia | 30 minutes after the block is performed
  The quality of the patient position will be assessed by Anesthesiologist B who administers spinal anesthesia and is blind to the blocks performed (0 = insufficient, 1 = sufficient, 2 = good, 3 = optimal)
The Necessity for Sedoanalgesia for Positional Pain in Unilateral Spinal Anesthesia | 30 minutes after the block is performed
  The necessity for sedoanalgesia for pain in the unilateral spinal anesthesia position will be assessed by the Anesthesiologist B who administers spinal anesthesia and is blind to the blocks performed. Rescue sedoanalgesia (propofol - ketamine combination) will be applied to patients with VAS >3. Patients will be recorded as 1 = needing sedoanalgesia, 2 = not needing sedoanalgesia.
Postoperative Pain | Postoperative 2nd, 6th, 12th and 24th hours
  Postoperative pain at 2nd, 6th, 12th and 24th hours will be evaluated using VAS by Anesthesiologist B who is blind to the blocks performed.
The Time Until First Opiod Requirement | Postoperative first 24-hour-period
  Within the first 24-hour-period, as soon as the VAS >3, intravenous opiod (1 mg/kg Tramadol) will be administered and time to first opioid requirement will be recorded.
Postoperative First 24-hour-period Total Opioid Consumption | Postoperative first 24-hour-period
  Total opioid (tramadol) consumption in the first 24 hours postoperatively will be recorded in mg/kg/day.
Patient and Surgeon Satisfaction | Immediately after the surgery
  Patient and surgeon satisfaction will be evaluated as: 1 = Complete dissatisfaction, 2 = Moderate dissatisfaction, 3 = Moderate satisfaction, 4 = Complete satisfaction
Undesirable Side Effects | Postoperative first 24-hour-period
  Recorded when there is vascular puncture, hematoma, signs of LA toxicity.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Bozyaka Training and Research Hospital, Izmir, Karabaglar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Hebbard P, Ivanusic J, Sha S. Ultrasound-guided supra-inguinal fascia iliaca block: a cadaveric evaluation of a novel approach. Anaesthesia. 2011 Apr;66(4):300-5. doi: 10.1111/j.1365-2044.2011.06628.x. Epub 2011 Feb 24. PMID 21401544
- [Background] Winnie AP, Ramamurthy S, Durrani Z. The inguinal paravascular technic of lumbar plexus anesthesia: the "3-in-1 block". Anesth Analg. 1973 Nov-Dec;52(6):989-96. No abstract available. PMID 4796576